CLINICAL TRIAL: NCT00841139
Title: Metabolic Manipulation in Chronic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Principal Investigator, Roger Beadle, Research Fellow to Professor MP Frenneaux, University Hospital Birmingham NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004-004965-14; MREC: 06/Q2707/7 (Other: Regional Ethics Committe); R&D Birminham: RRK 2785 (Other: Hospital R&D); MHRA: 21761/0003/001 (Other: MHRA); 2004-004965-14 (EudraCT Number)
Record Dates: First submitted 2009-02-06; First posted 2009-02-11 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Chronic Heart Failure
Keywords: perhexiline; idiopathic dilated cardiomyopathy; magnetic resonance spectroscopy; cardiac energetics
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — Perhexiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perhexiline (Experimental): perhexiline 100mg bd for 1 month duration
  Interventions: Drug: Perhexiline
- Placebo (Placebo Comparator): placebo one tablet bd for 1 month duration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Perhexiline — 100mg o bd
  Other Names: Pexsig
  Arms: Perhexiline
Drug: Placebo — 1 tablet bd
  Arms: Placebo

SUMMARY:
Conventional measures used for the treatment of chronic heart failure act predominantly by reducing the work performed by the heart. In a recent study, the investigators showed that one drug (perhexiline) substantially improved symptoms and cardiac function in heart failure. The investigators wish to confirm these findings and test whether or not this drug acts by altering the heart's energy source thus augmenting the energetic status and work efficiency of the heart.

DETAILED DESCRIPTION:
Perhexiline maleate is an antianginal agent which increases the efficiency of energy production by shifting substrate utilisation from free fatty acids towards glucose. We showed that perhexiline therapy was highly effective in improving exercise capacity, symptoms and cardiac function in patients with systolic heart failure of both ischaemic and non ischaemic aetiology. Perhexiline acts by inhibiting both carnitine palmitoyl transferase-1 (CPT-1) and CPT-2, which are key enzymes in mitochondrial free fatty acid uptake. This leads to increased myocardial glucose substrate utilization. Further we wish to ascertain whether or not this drug improves cardiac energetics and efficiency by altering substrate utilization. In this proposal we will assess the cardiac function (by cardiac Magnetic Resonance Imaging MRI), cardiac energetic status (by cardiac Magnetic Resonance Spectroscopy MRS), cardiac efficiency (via pressure-volume loops) and substrate utilization (via left and right heart catheterization), following one month of perhexiline therapy or placebo in patients with symptomatic idiopathic dilated cardiomyopathy on optimal conventional heart failure medications. An interim analysis is planned after 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Optimally-medicated idiopathic dilated cardiomyopathy
* Symptomatic ( NYHA IIb-III)
* Impaired left ventricular systolic function (EF < 40%)

Exclusion Criteria:

* Abnormal liver function tests (defined as above twice the upper limit of normal (ULN))
* Concomitant use of Amiodarone , Quinidine , Haloperidol or Selective serotonin (5HT) uptake inhibitors such as Fluoxetine and Paroxetine which may inhibit the CYP2D6 enzyme.
* Pre-existing evidence of peripheral neuropathy.
* Women of childbearing potential.
* Patients with implantable cardiac devices (or any other contraindication to MRI).
* Obesity ( BMI > 32)
* Obstructive sleep apnea syndrome
* Patients with known hypersensitivity to perhexiline
* Patients with impaired renal function (Creatinine > 250 µmol/L)
* Valvular heart disease defined as more than moderate valvular stenosis or regurgitation.
* Atrial Fibrillation

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in cardiac energetics as demonstrated by resting myocardial PCr/ATP ratio from cardiac MRS | 1 Month

SECONDARY OUTCOMES:
Change in mechanical efficiency (external work / MVO2) | 1 Month
Change in respiratory quotient | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Frenneaux, MBBS MD, Principal Investigator — University of Birmingham; Roger M Beadle, MBBS, Study Director — University of Birmingham
Locations (2):
- United Kingdom (2):
  - University Hospitals Brimingham NHS Foundation Trust, Birmingham, West Midlands
  - University of Birmingham, Birmingham, West Midlands

REFERENCES:
- [Derived] Beadle RM, Williams LK, Kuehl M, Bowater S, Abozguia K, Leyva F, Yousef Z, Wagenmakers AJ, Thies F, Horowitz J, Frenneaux MP. Improvement in cardiac energetics by perhexiline in heart failure due to dilated cardiomyopathy. JACC Heart Fail. 2015 Mar;3(3):202-11. doi: 10.1016/j.jchf.2014.09.009. Epub 2015 Jan 28. PMID 25650370
- [Derived] Beadle RM, Williams LK, Abozguia K, Patel K, Leon FL, Yousef Z, Wagenmakers A, Frenneaux MP. Metabolic manipulation in chronic heart failure: study protocol for a randomised controlled trial. Trials. 2011 Jun 6;12:140. doi: 10.1186/1745-6215-12-140. PMID 21645332